CLINICAL TRIAL: NCT06509100
Title: Altitudes: A Blended Digital Health Intervention to Support Caregivers and Other Supporters of Young People With Psychosis
Brief Title: Altitudes: A Digital Intervention to Support Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Department of Health and Human Services (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 24-1141
Record Dates: First submitted 2024-07-09; First posted 2024-07-19 (Actual); Results first posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-10

CONDITIONS: Care Burden; Care Giving Burden; Caregiver Burnout; Caregiver Stress; Caregiver Wellbeing; Support, Family
Keywords: Digital Intervention; Social Media; Virtual Therapeutic Content; Virtual Educational Content; Supporters; Caregiving
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Altitudes Condition (Experimental): Individuals whose loved ones are experiencing first-episode psychosis (FEP) and receiving services from OASIS, SHORE, Eagle, Encompass, AEGIS, and WeCare2), STEP programs, or community services will be recruited to participate in a digital platform, Altitudes, for 6 months as part of an adjunct service to the clinic's services. Participants will have access to and encouraged to use the educational and therapeutic content as well as the moderated online community network during their time engaging with the platform. They will be asked to complete a battery of measures at baseline, 3-months, and 6 months.
  Interventions: Device: Device: Altitudes USA

INTERVENTIONS:
Device: Device: Altitudes USA — Experimental participants will be onboarded to the digital platform, including the different spaces and how to use the site. The site includes educational and therapeutic content that is tailored to each individual and their current needs and experiences, including psychoeducation, supporting their loved one, self- care, social support, and so on. Further, the platform includes a moderated social media function, where users and family peer workers can post text, images, videos, and comments to connect and share their experiences. The site is monitored by graduated students and trained clinicians.

SUMMARY:
The purpose of the present study is to investigate the feasibility, accessibility, and potential clinical benefits of implementing a moderated online social media platform with therapeutic content, Altitudes, to parents, caregivers, and supporters of young people with psychosis across the state of North Carolina, including in Coordinated Specialty Care (CSC) programs, Specialized Treatment Early in Psychosis (STEP) programs, and other community services where caregivers or supporters of young persons experiencing psychosis receive care. The investigators will evaluate acceptability and feasibility with up to 50 caregivers and supporters over the course of 6 months. Acceptability and usability will be assessed with various acceptability measures with the Altitudes caregivers and supporters, and caregivers and supporters' engagement with the digital platform. The investigators will additionally evaluate the impact of the platform on caregiver and supporter's psychological status, well-being, and social support, as measured via self-report questionnaires.

DETAILED DESCRIPTION:
Purpose: The purpose of the present study is to investigate the feasibility, accessibility, and potential clinical benefits of implementing a moderated online social media platform with therapeutic content, Altitudes, to parents, caregivers, and supporters of young people with psychosis across the state of North Carolina, including in CSC programs, STEP programs, and other community services where caregivers or supporters of young persons experiencing psychosis receive care.

Participants: Fifty parent or supporter participants from CSC clinics (OASIS, SHORE, Eagle, Encompass, AEGIS, and WeCare2), STEP programs, or community services will be recruited for Altitudes.

Procedures (methods): All participants will be recruited over a 20-week to 28-week period at from the North Carolina's community services. Participants will engaged with the digital platform, known as Altitudes, for approximately 6 months. Site usage information as well as feedback about their experience will be collected from these participants through the Altitudes platform. Site usage information (e.g., number of posts/comments made on the site, the number and types of 'Journeys' or 'Tracks' [psychoeducation and therapeutic content] completed by participants, etc.) will be collected automatically through the Altitudes platform. Before being given access to Altitudes, a research coordinator, family peer support specialist, or moderator will provide instructions and guidance for using the site (i.e., Altitudes onboarding). Experiences, wellbeing, and support measures will be collected at baseline, mid-treatment (~3 months) and post-treatment (~6 months) for the Altitudes participants. As Altitudes involves psychoeducational and therapeutic content, this platform is considered an adjunct to care parents and supporters may be receiving. As such, Altitudes participants will not be compensated for their involvement in the platform. Site usage information will be collected automatically through the Altitudes site. However, Altitudes participants will be compensated for providing feedback about their experience with Altitudes as well as for completing other assessments. Finally, Altitudes will be monitored at least once daily by trained family peer support specialists, master's or Ph.D. level clinicians, and/or graduate students with relevant clinical/research experience with individuals experiencing psychosis and their supporters. Dr. Emily Parsons, trained clinical psychologist and family therapist, will lead bi-weekly supervision calls to ensure appropriate care and support of Altitudes participants involved in this project, to discuss case conceptualization and suggestions for engaging individuals in the platform, as well as to monitor any potential safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* The participants must be a parent, caregiver, or supporter of a young person who is currently receiving treatment from a CSC program for FEP or STEP clinic, on the waitlist to receive services from the CSC, who has recently graduated/discharged from a CSC program, or was referred to the study from the community (via Early Psychosis Interventions of North Carolina (EPI-NC) warm line, community psychiatrist/therapist, or inpatient/outpatient mental health services) where young person is experiencing psychosis but was not referred or enrolled in CSC
* Parent, caregiver, or supporter must be > 18 years of age
* Participants recruited from NC CSC programs (i.e., OASIS, SHORE, Encompass, Eagle, AEGIS, WeCare2), STEP programs, and the community screening process
* Parent, caregiver, or supporter must have access to internet through a mobile phone, tablet, or computer

Exclusion Criteria:

* Parent or caregiver is currently engaged in legal action against the loved one experiencing psychosis
* Parent or caregiver does not speak and understand English as the platform, its moderation, interviews, and measures are available only in English
* Parent, caregiver, or supporter is <18 years of age

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2024-09-03 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelsey R Ludwig, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Diana Perkins, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication and provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with University of North Carolina (UNC).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 9 and continuing for 36 months following publication
Access Criteria: Requesting investigator has appropriate approval (see above) and an executed data use/sharing agreement with UNC.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Altitudes Condition
Started | 17
Completed | 15
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Altitudes Condition
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.529 (8.718)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 3
  Female | 14
  Non-binary | 0
  Transgender female | 0
  Transgender male | 0
  Other (please specify) | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Altitudes Health Care Climate Questionnaire (A-HCCQ) - Total Score
Description: The Altitudes Health Care Climate Questionnaire is a 15-item scale. Answers are on a 7-point Likert scale (1-7) with options "Strongly Disagree", "Mildly Disagree", "Slightly Disagree", "Neutral", "Slightly Agree", "Mildly Agree", and "Strongly Agree". Possible scores range from 15 to 105 with higher scores reflecting better perceptions of their relationship with Altitudes moderators.
Time Frame: [Time Frame: Month 3, Month 6]
Population: Data are only reported for participants who completed both mid-treatment and post treatment assessments.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Altitudes Condition
Number analyzed (Participants) | 11
Scores on a scale | 0.091 (16.257)

2. Primary Outcome: Mean Change in Working Alliance Inventory for Guided Internet Interventions (WAI-I) - Total Score
Description: The Working Alliance Inventory for Guided Internet Interventions (WAI-I) is a 12-item scale. Answers are on a 5-point scale with options "seldom", "sometimes", "fairly often", "very often", and "always". Possible scores are averaged across items and range from 1 to 5. Higher scores indicate greater therapeutic alliance.
Time Frame: [Time Frame: Month 3, Month 6]
Population: Data are only reported for participants who completed both mid-treatment and post treatment assessments.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Altitudes Condition
Number analyzed (Participants) | 11
Scores on a scale | 1.091 (7.529)

3. Primary Outcome: Mean Change in Working Alliance Inventory for Guided Internet Interventions (WAI-I) - Task and Goals Subscale
Description: The Working Alliance Inventory for Guided Internet Interventions (WAI-I) task and goals subscale is an 8-item scale. Answers are on a 5-point scale with options "seldom", "sometimes", "fairly often", "very often", and "always". Possible scores are averaged across items and range from 1 to 5. Higher scores indicate greater agreement between the therapist and client on tasks and goals.
Time Frame: [Time Frame: Month 3, Month 6]
Population: Data are only reported for participants who completed both mid-treatment and post treatment assessments.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Altitudes Condition
Number analyzed (Participants) | 11
Scores on a scale | 0.273 (6.680)

4. Primary Outcome: Mean Change in Working Alliance Inventory for Guided Internet Interventions (WAI-I) - Bond Subscale
Description: The Working Alliance Inventory for Guided Internet Interventions (WAI-I) is a 4-item scale. Answers are on a 5-point scale with options "seldom", "sometimes", "fairly often", "very often", and "always". Possible scores are averaged across items and range from 1 to 5. Higher scores indicate stronger bond with the supporting therapist.
Time Frame: [Time Frame: Month 3, Month 6]
Population: Data are only reported for participants who completed both mid-treatment and post treatment assessments.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Altitudes Condition
Number analyzed (Participants) | 11
Scores on a scale | 0.818 (1.722)

5. Primary Outcome: Mean Change in Altitudes Perceived Competence Scale (A-PCS) - Total Score
Description: The Altitudes Health Care Climate Questionnaire is a 4-item scale. Answers are on a 7-point Likert scale with options "Not at all true"[1], "Somewhat true"[4], "Very true"[7] with a sliding scale between answers. Possible scores range from 4 to 28. Higher scores indicate stronger perceived competence and ability in using the Altitudes platform.
Time Frame: [Time Frame: Month 3, Month 6]
Population: Data are only reported for participants who completed both mid-treatment and post treatment assessments.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Altitudes Condition
Number analyzed (Participants) | 11
Scores on a scale | -0.545 (2.067)

6. Primary Outcome: Mean Change in Altitudes Usability Questionnaire (AUQ) - Overall Impressions of Platform Subscale
Description: The Altitudes Health Care Climate Questionnaire is a 20-item scale. The overall impressions of the platform scale is three 7-point Likert scale answers with options of "Strongly Disagree", "Mildly Disagree", "Slightly Disagree", "Neutral", "Slightly Agree", "Mildly Agree", and "Strongly Agree". Possible scores range from 3 to 21. Higher scores indicate better overall impressions of the Altitudes platform.
Time Frame: [Time Frame: Month 3, Month 6]
Population: Data are only reported for participants who completed both mid-treatment and post treatment assessments.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Altitudes Condition
Number analyzed (Participants) | 11
Scores on a scale | 0.455 (2.296)

7. Primary Outcome: Mean Change in Altitudes Usability Questionnaire (AUQ) - Perception of Other Platform Users Subscale
Description: The Altitudes Health Care Climate Questionnaire is a 20-item scale. The perception of other platform users subscale is four 7-point Likert scale answers with options of "Strongly Disagree", "Mildly Disagree", "Slightly Disagree", "Neutral", "Slightly Agree", "Mildly Agree", and "Strongly Agree". Possible scores range from 4 to 28. Higher scores indicate better perception of interactions with other Altitudes participants.
Time Frame: [Time Frame: Month 3, Month 6]
Population: Data are only reported for participants who completed both mid-treatment and post treatment assessments.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Altitudes Condition
Number analyzed (Participants) | 11
Scores on a scale | -0.182 (2.822)

8. Primary Outcome: Mean Change in Altitudes Usability Questionnaire (AUQ) - Safety and Confidentiality Subscale
Description: The Altitudes Health Care Climate Questionnaire is a 20-item scale. The safety and confidentiality subscale is two 7-point Likert scale answers with options of "Strongly Disagree", "Mildly Disagree", "Slightly Disagree", "Neutral", "Slightly Agree", "Mildly Agree", and "Strongly Agree". Possible scores range from 2 to 14. Higher scores indicate higher perceived safety and confidentiality when using the platform.
Time Frame: [Time Frame: Month 3, Month 6]
Population: Data are only reported for participants who completed both mid-treatment and post treatment assessments.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Altitudes Condition
Number analyzed (Participants) | 11
Scores on a scale | -0.182 (2.786)

9. Primary Outcome: Mean Change in Altitudes Usability Questionnaire (AUQ) - Moderation and Peer Support Subscale
Description: The Altitudes Health Care Climate Questionnaire is a 20-item scale. The moderation and peer support subscale is three 7-point Likert scale answers with options of "Strongly Disagree", "Mildly Disagree", "Slightly Disagree", "Neutral", "Slightly Agree", "Mildly Agree", and "Strongly Agree". Possible scores range from 3 to 21. Higher scores indicate higher regard of the moderators and peer support on the Altitudes platform.
Time Frame: [Time Frame: Month 3, Month 6]
Population: Data are only reported for participants who completed both mid-treatment and post treatment assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition
Number analyzed (Participants) | 11
score on a scale | -0.455 (3.267)

10. Primary Outcome: Mean Change in Altitudes Usability Questionnaire (AUQ) - Ideas for Increased Engagement Subscale
Description: The Altitudes Health Care Climate Questionnaire is a 20-item scale. The ideas for increased engagement subscale is five 7-point Likert scale answers with options of "Strongly Disagree", "Mildly Disagree", "Slightly Disagree", "Neutral", "Slightly Agree", "Mildly Agree", and "Strongly Agree". Possible scores range from 5 to 35. Each question has to be interrupted individually to assess of the subscale.
Time Frame: [Time Frame: Month 3, Month 6]
Population: Data are only reported for participants who completed both mid-treatment and post treatment assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition
Number analyzed (Participants) | 11
score on a scale | 0.182 (2.960)

11. Primary Outcome: Mean Change in Altitudes Usability Questionnaire (AUQ) - Barriers to Use Subscale
Description: The Altitudes Health Care Climate Questionnaire is a 20-item scale. The barriers to use subscale is six 7-point Likert scale answers with options of "Strongly Disagree", "Mildly Disagree", "Slightly Disagree", "Neutral", "Slightly Agree", "Mildly Agree", and "Strongly Agree". Possible scores range from 6 to 42. Lower scores indicate less issues with barriers to engaging with the platform.
Time Frame: [Time Frame: Month 3, Month 6]
Population: Data are only reported for participants who completed both mid-treatment and post treatment assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition
Number analyzed (Participants) | 11
score on a scale | 1.818 (2.562)

12. Primary Outcome: Mean Engagement With the Altitudes Platform
Description: The Altitudes platform passively collects engagement data, including the number of therapy material accessed, number of problem-solving discussion forums (i.e., "talk-it-outs"), and any posts, comments, or reactions (emojis to other users' posts/comments) made on the platform. The investigators will provide the means and standard deviations for these site usage categories throughout the study period.
Time Frame: [Up to Month 6]
Measure: Mean (Standard Deviation); unit: clicks per category
Arm/Group | Altitudes Condition
Number analyzed (Participants) | 17
clicks per category
  Talk-it-out | 0.12 (0.332)
  Posts on community page | 1.71 (2.201)
  Reactions on community page | 7.35 (9.893)
  Comments on community page | 3.12 (6.214)
  Therapy | 41.41 (52.571)

13. Secondary Outcome: Mean Change in Medical Outcomes Study (MOS) Social Support Survey - Total Score
Description: The MOS Social Support Survey is a 19-item scale. Answers are on a 5-point scale with options "none of the time", "a little of the time", "some of the time", "most of the time", and "all of the time". Possible scores range from 19 to 95. Higher scores reflect higher feelings of social support (more perceived social support). The MOS Social Support Survey is a part of the PhenX Toolkit.
Time Frame: [Time Frame: Baseline, Up to Month 6]
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition
Number analyzed (Participants) | 17
score on a scale | 1.353 (16.159)

14. Secondary Outcome: Mean Change in Generalized Anxiety Disorder 7-item (GAD-7) - Total Score
Description: The GAD-7 is an 7-item scale. Answers are on a 4-point scale (0 = not at all; 3 = nearly every day) Possible scores range from 0 to 21. Higher scores reflect worse anxiety).
Time Frame: [Time Frame: Baseline, Up to Month 6]
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition
Number analyzed (Participants) | 17
score on a scale | -0.588 (5.075)

15. Secondary Outcome: Mean Change in Patient Health Questionnaire (PHQ) - Total Score
Description: The PHQ is an 8-item scale. Answers are on a 4-point scale (0 = not at all; 3 = nearly every day). Possible scores range from 0 to 24. Higher scores reflect a greater severity of depression.
Time Frame: [Time Frame: Baseline, Up to Month 6]
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition
Number analyzed (Participants) | 17
score on a scale | -1.118 (5.476)

16. Secondary Outcome: Mean Change in Five Facet Mindfulness Questionnaire: 24-item (FFMQ-24) - Non-Reactivity Subscale
Description: The Five Facet Mindfulness Questionnaire: 24 is a 24-item self-report questionnaire designed to measure an individual's mindful self-awareness. The non-reactivity subscale is 5 items with answers are on a 5-point Likert scale of "Never or very rarely true", "Rarely true", "Sometimes true", "Often true", and "Very often true or always true". Possible scores range from 5 to 25 with higher scores indicate more mindful non-reactivity to thoughts and feelings.
Time Frame: [Time Frame: Baseline, Up to Month 6]
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition
Number analyzed (Participants) | 17
score on a scale | 0.294 (1.863)

17. Secondary Outcome: Mean Change in Five Facet Mindfulness Questionnaire: 24-item (FFMQ-24) - Non-Judgmental Inner Experience Subscale
Description: The Five Facet Mindfulness Questionnaire: 24 is a 24-item self-report questionnaire designed to measure an individual's mindful self-awareness. The non-judgemental subscale is 5 items with answers are on a 5-point Likert scale of "Never or very rarely true", "Rarely true", "Sometimes true", "Often true", and "Very often true or always true". Possible scores range from 5 to 25 once appropriate items have been reversed scored with higher scores indicate more nonjudgmental thoughts towards their beliefs and feelings.
Time Frame: [Time Frame: Baseline, Up to Month 6]
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition
Number analyzed (Participants) | 17
score on a scale | 0.235 (1.985)

18. Secondary Outcome: Mean Change in Five Facet Mindfulness Questionnaire: 24-item (FFMQ-24) - Mindful Action Subscale
Description: The Five Facet Mindfulness Questionnaire: 24 is a 24-item self-report questionnaire designed to measure an individual's mindful self-awareness. The mindful action subscale is 5 items with answers are on a 5-point Likert scale of "Never or very rarely true", "Rarely true", "Sometimes true", "Often true", and "Very often true or always true". Possible scores range from 5 to 25 after appropriate items have been reversed scored with higher scores indicate more awareness around their actions and experiences.
Time Frame: [Time Frame: Baseline, Up to Month 6]
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition
Number analyzed (Participants) | 17
score on a scale | -0.059 (2.410)

19. Secondary Outcome: Mean Change in Five Facet Mindfulness Questionnaire: 24-item (FFMQ-24) - Description Subscale
Description: The Five Facet Mindfulness Questionnaire: 24 is a 24-item self-report questionnaire designed to measure an individual's mindful self-awareness. The description subscale is 5 items with answers are on a 5-point Likert scale of "Never or very rarely true", "Rarely true", "Sometimes true", "Often true", and "Very often true or always true". Possible scores range from 5 to 25 after reverse scoring of appropriate items with higher scores indicate more to describe their feelings and experiences.
Time Frame: [Time Frame: Baseline, Up to Month 6]
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition
Number analyzed (Participants) | 17
score on a scale | 0.588 (1.278)

20. Secondary Outcome: Mean Change in Five Facet Mindfulness Questionnaire: 24-item (FFMQ-24) - Observation Subscale
Description: The Five Facet Mindfulness Questionnaire: 24 is a 24-item self-report questionnaire designed to measure an individual's mindful self-awareness. The observation subscale is 3 items with answers are on a 5-point Likert scale of "Never or very rarely true", "Rarely true", "Sometimes true", "Often true", and "Very often true or always true". Possible scores range from 3 to 15 with higher scores indicate more observational awareness.
Time Frame: [Time Frame: Baseline, Up to Month 6]
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition
Number analyzed (Participants) | 17
score on a scale | 0.882 (1.691)

21. Secondary Outcome: Mean Change in Five Facet Mindfulness Questionnaire: 24-item (FFMQ-24) - Total Score
Description: The Five Facet Mindfulness Questionnaire: 24-item is a 24-item self-report questionnaire designed to measure an individual's mindful self-awareness. It can be divided into five subscales: Observing, Describing, Acting in Awareness, Non-judging, and Non-reactivity. Answers are on a 5-point Likert scale of "Never or very rarely true", "Rarely true", "Sometimes true", "Often true", and "Very often true or always true". Possible scores range from 24 to 120 once necessary questions (i.e., negative) have been reversed scored. Higher scores indicate more mindfulness and self- awareness.
Time Frame: [Time Frame: Baseline, Up to Month 6]
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition
Number analyzed (Participants) | 17
score on a scale | 2.059 (3.960)

22. Secondary Outcome: Mean Change in Self-Compassion Scale: Short Form (SCS) - Total Score
Description: The Self-Compassion Scale is a 12-item self-report questionnaire designed to measure an individual's self-compassion towards themselves as well as their feelings and emotions. It can be divided into six subscales with two questions for each: Self-Kindness, Self-Judgment, Common Humanity, Isolation, Mindfulness, Over-identified. Answers are on a 5- point scale ranging from 1 "Almost never" to 5 "Almost always." Total score is calculated by totaling the mean of each subscales and reversing the negative subscales (self-judgment, isolation, and over-identification) then taking the mean of the summed subscales. Possible scores range from 1 to 5 with higher scores indicate increased self-compassion.
Time Frame: [Time Frame: Baseline, Up to Month 6]
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition
Number analyzed (Participants) | 17
score on a scale | 0.064 (0.266)

23. Secondary Outcome: Mean Change in the Modified Psychosis Attitude Survey - Total Score
Description: The Modified Psychosis Attitudes Survey is a 19-item self-report questionnaire designed to measure an individual's beliefs and attitude towards psychosis (e.g., identifying psychosis, interacting with individuals experiencing psychosis, etc.). The survey can be divided into 4 subscales: perceived confidence, optimism, fulfillment, and stress-vulnerability orientation. Answers range from "Very strongly disagree", "Strongly disagree", "Mildly disagree", "Neutral", "Mildly agree", "Strongly agree", "Very strongly agree". Total score is obtained with summing each question, after reverse scoring appropriate questions. Possible scores range from 19 to 133. Higher total score indicates an increased knowledge, optimism, and attitudes towards psychosis.
Time Frame: [Time Frame: Baseline, Up to Month 6]
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Altitudes Condition
Number analyzed (Participants) | 17
score on a scale | 3.353 (8.817)

24. Secondary Outcome: Mean Change in University of California, Los Angeles (UCLA) Loneliness Scale - Total Score
Description: The UCLA Loneliness scale is a 20-item scale. Answers are on a 4-point scale with options "I often feel this way," "I sometimes feel this way," "I rarely feel this way," and "I never feel this way." Possible scores range from 20 to 80. Higher scores reflect worse outcomes (greater feelings of loneliness). The UCLA Loneliness Scale is a part of the PhenX Toolkit.
Time Frame: [Time Frame: Baseline, up to Month 6]
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition
Number analyzed (Participants) | 17
score on a scale | -2.588 (3.675)

25. Secondary Outcome: Mean Change in the Brief Coping Orientation to Problems Experienced (COPE) Scale - Emotion-Focused Subscale
Description: The Brief-COPE is a 28-item self-report questionnaire designed to measure effective and ineffective ways to cope with a stressful life event. The emotion-focused subscale is 12 items. Answers are on a 4-point scale ranging from 1 "I haven't been doing this at all" to 4 "I have been doing this a lot." Possible scores range from 12 to 48. Higher scores on each reflect more frequent use of emotion focused coping.
Time Frame: [Time Frame: Baseline, Up to Month 6]
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition
Number analyzed (Participants) | 17
score on a scale | 0.706 (6.302)

26. Secondary Outcome: Mean Change in the Brief Coping Orientation to Problems Experienced (COPE) Scale - Avoidant-Focused Subscale
Description: The Brief-COPE is a 28-item self-report questionnaire designed to measure effective and ineffective ways to cope with a stressful life event. The avoidant-focused subscale is 8 items. Answers are on a 4-point scale ranging from 1 "I haven't been doing this at all" to 4 "I have been doing this a lot." Possible scores range from 8 to 32. Higher scores on each reflect more frequent use of avoidance for coping.
Time Frame: [Time Frame: Baseline, Up to Month 6]
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition
Number analyzed (Participants) | 17
score on a scale | -0.471 (5.026)

27. Secondary Outcome: Mean Change in the Brief Coping Orientation to Problems Experienced (COPE) Scale - Problem-Focused Subscale
Description: The Brief-COPE is a 28-item self-report questionnaire designed to measure effective and ineffective ways to cope with a stressful life event. The problem-focused subscale is 8 items. Answers are on a 4-point scale ranging from 1 "I haven't been doing this at all" to 4 "I have been doing this a lot." Possible scores range from 8 to 32. Higher scores on each reflect more frequent use of problem focused coping.
Time Frame: [Time Frame: Baseline, Up to Month 6]
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition
Number analyzed (Participants) | 17
score on a scale | 0.059 (3.665)

28. Secondary Outcome: Mean Change in Family Questionnaire of Expressed Emotion - Emotional Overinvolvement (EOI) Subscale
Description: The Family Questionnaire (FQ) is a 20-item, self-administered questionnaire that measures expressed emotion status (criticism and emotional over involvement (EOI)) of family members toward patients with mental illness. The EOI subscale consists of 10 items with each item is rated on a 4-point scale (1 = never/very rarely; 4 = very often). The EOI subscale is scored by adding together the ratings from the individual items. Possible scores ranging from 10 to 40 with higher scores indicating greater levels of emotional overinvolvement with their loved one.
Time Frame: [Time Frame: Baseline, Up to Month 6]
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition
Number analyzed (Participants) | 17
score on a scale | -2.353 (4.344)

29. Secondary Outcome: Mean Change in Family Questionnaire of Expressed Emotion - Critical Comments Subscale
Description: The Family Questionnaire (FQ) is a 20-item, self-administered questionnaire that measures expressed emotion status (criticism and emotional over involvement (EOI)) of family members toward patients with mental illness. The subscale is 10-items and is rated on a 4-point scale (1 = never/very rarely; 4 = very often). It is scored by adding together the ratings from the individual items. Possible scores ranging from 10 to 40 with higher scores indicating greater levels of critical comments with their loved one.
Time Frame: [Time Frame: Baseline, Up to Month 6]
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition
Number analyzed (Participants) | 17
score on a scale | -1.294 (4.972)

30. Secondary Outcome: Mean Change in Family Questionnaire of Expressed Emotion - Total Score
Description: The Family Questionnaire (FQ) is a 20-item, self-administered questionnaire that measures expressed emotion status (criticism and emotional over involvement (EOI)) of family members toward patients with mental illness. The FQ has two subscales: critical comments, and EOI. Each item is rated on a 4-point scale (1 = never/very rarely; 4 = very often). The FQ is scored by adding together the ratings from the individual items. Possible scores range from 20 to 80 with higher scores indicating greater levels of expressed emotion.
Time Frame: [Time Frame: Baseline, Up to Month 6]
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition
Number analyzed (Participants) | 17
score on a scale | -3.647 (8.276)

31. Secondary Outcome: Mean Change in the Experience of Caregiving Inventory (ECI) - Negative Experiences Subscale
Description: The ECI Scale is a 66-item scale. Answers are on a 5-point scale starting at 0 with options "never," "rarely," "sometimes," "often," and "nearly always". The negative experience subscale is 52 items with possible scores range from 0 to 208. Higher scores reflect feeling less prepared to provide caregiving and more negative experiences in caregiving.
Time Frame: [Time Frame: Baseline, Up to Month 6]
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition
Number analyzed (Participants) | 17
score on a scale | -10.824 (18.822)

32. Secondary Outcome: Mean Change in the Experience of Caregiving Inventory (ECI) - Positive Experience Subscales
Description: The ECI Scale is a 66-item scale. Answers are on a 5-point scale starting at 0 with options "never," "rarely," "sometimes," "often," and "nearly always". The positive experience subscale is 14 items with possible scores range from 0 to 56. Higher scores indicate greater feelings of preparedness and experiences with caregiving.
Time Frame: [Time Frame: Baseline, Up to Month 6]
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition
Number analyzed (Participants) | 17
score on a scale | 4.059 (4.930)

33. Other Pre Specified Outcome: Mean Change in the PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 (PCL-5)
Description: The PCL-5 is a 20-item self-report measure of the 20 DSM-5 symptoms of Post Traumatic Stress Disorder (PTSD). Included in the scale are four domains consistent with the four criteria of PTSD in DSM-5: Re-experiencing (criterion B), Avoidance (criterion C), Negative alterations in cognition and mood (criterion D), and Hyper-arousal (criterion E). Answers are on a 5-point scale including "Not at all," "A little bit," "Moderately," "Quite a bit," and "Extremely" and with total scores ranging from 0 to 80. Higher scores on the PCL-5 reflect more severe trauma-related symptoms.
Time Frame: [Time Frame: Baseline, Up to Month 6]
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Altitudes Condition
Number analyzed (Participants) | 17
score on a scale | -2.647 (7.348)

ADVERSE EVENTS:
Time Frame: From Baseline to end of follow-up, up to 6 months.
Arm/Group | Altitudes Condition
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-18): https://cdn.clinicaltrials.gov/large-docs/00/NCT06509100/Prot_SAP_000.pdf
  • Informed Consent Form (2024-05-28): https://cdn.clinicaltrials.gov/large-docs/00/NCT06509100/ICF_001.pdf